CLINICAL TRIAL: NCT05055401
Title: The Proficiency and Efficiency of Airway Management Skills Amongst Anesthesia Providers: A Multicenter Baseline Assessment
Brief Title: Airway Management Skills Amongst Anesthesia Providers
Status: Enrolling by invitation | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104249
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Airway Management
Keywords: Airway Management; Intubation; High Fidelity Mannikin; Anesthesia Providers
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anesthesiology providers: Group will contain anesthesiologists, CRNA and AAs. The type of healthcare professional participating will be recorded along with the years of experience the participant has. Each participants experience will be categorized into three ranges, 0-3 years, 3-10 years, and 10+ years of experience. For further clarification and analysis, the healthcare professional's normal practice setting will also be recorded including inpatient, outpatient, or hybrid (inpatient and outpatient) settings. All providers will be analyzed together.
  Interventions: Procedure: Direct Laryngoscopy; Procedure: Laryngeal Mask Airways; Procedure: Video Laryngoscopy

INTERVENTIONS:
Procedure: Direct Laryngoscopy — The participant will perform a direct laryngoscopy on a Laerdal SimMan 3G under healthy conditions and under limited cervical range of motion.
Procedure: Laryngeal Mask Airways — The participant will perform LMA placement on a Laerdal SimMan 3G under healthy conditions and under full tongue edema.
Procedure: Video Laryngoscopy — The participant will perform video laryngoscopy on a Laerdal SimMan 3G under healthy conditions and under half tongue edema with pharyngeal obstruction.

SUMMARY:
The aim of this study is to evaluate the efficiency and proficiency of three common airway management techniques amongst among anesthesia providers who maintain airway management privileges in our health system.

DETAILED DESCRIPTION:
Airway management may take place in a variety of settings with varying degrees of urgency, ranging from performance for elective operative procedures to life-threatening emergencies. An appropriate psychomotor skill set is needed to perform the procedures utilized for airway management, and the time required to do so may impact patient outcomes. Prolonged periods of apnea and accompanying hypoxia can lead to brain damage or death. This research is designed to evaluate the proficiency of anesthesia providers who are responsible for practicing airway management in hospitals or health systems in the United States, including Anesthesiologists, Certified Registered Nurse Anesthetists, and Anesthesiology Assistants. We are attempting to establish a baseline level of proficiency by quantifying the time it takes to achieve successful airway management and the number of attempts required to do so utilizing a high fidelity manikin programmed to simulate various physiological conditions. This baseline information could then be used to manage the decisions made by hospitals or health systems related to airway management in the future, or to redefine the policies and procedures established for performing these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant
* Participants are presently employed as an anesthesiologist (previously completed an anesthesiology residency), CRNA or AA at a participating institution
* Participants have active airway management privileges with their institution

Exclusion Criteria:

* Participants are not employed by their institution
* Refusal of the participant to sign a consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All employees of the respective anesthesia departments employed by Prisma Health will be offered participation in this study including: anesthesiologists (previously completed anesthesiology residency), certified registered nurse anesthetists (CRNA), and anesthesia assistants (AA).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of Attempts to Achieve Successful Airway Management | Immediate Post-Procedure
  A successful attempt for any of the three procedures will be documented when a participant attaches a bag/valve and attempts a ventilation resulting in the presence of end-tidal carbon dioxide (which will be displayed when the device is properly placed). Failed attempts for any of the three procedures will be documented when a participant attaches a bag/valve device and attempts ventilation for purposes of confirming the presence of end-tidal carbon dioxide (which will not be displayed if the device is improperly placed). Three sequential failed attempts will result in a failure to achieve successful airway management.
Time Required to Achieve Successful Airway Management | Immediate Post-Procedure
  Time will be measured manually via stopwatch. Time measurement for all three procedures will begin when the participant picks up the laryngoscope, video laryngoscope, or LMA having signaled his/her intention to begin the procedure. Time measurement will end upon detection of end-tidal carbon dioxide by the mannikin as evidenced on a standard patient monitor connected to the mannikin for this purpose. Time measurement will continue during failed attempts and subsequent efforts to successfully perform the procedure. Time measurement will be stopped upon successful end-tidal carbon dioxide measurement, three sequential failed attempts to perform a procedure, or after a total of five minutes have passed.

CONTACTS AND LOCATIONS:
Overall Officials: Robert R. Morgan, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambrosio A, Pfannenstiel T, Bach K, Cornelissen C, Gaconnet C, Brigger MT. Difficult airway management for novice physicians: a randomized trial comparing direct and video-assisted laryngoscopy. Otolaryngol Head Neck Surg. 2014 May;150(5):775-8. doi: 10.1177/0194599814521380. Epub 2014 Jan 29. PMID 24477825
- [Background] Bhattacharjee S, Maitra S, Baidya DK. A comparison between video laryngoscopy and direct laryngoscopy for endotracheal intubation in the emergency department: A meta-analysis of randomized controlled trials. J Clin Anesth. 2018 Jun;47:21-26. doi: 10.1016/j.jclinane.2018.03.006. Epub 2018 Mar 14. PMID 29549828
- [Background] Bucx MJ, van Geel RT, Wegener JT, Robers C, Stijnen T. Does experience influence the forces exerted on maxillary incisors during laryngoscopy? A manikin study using the Macintosh laryngoscope. Can J Anaesth. 1995 Feb;42(2):144-9. doi: 10.1007/BF03028268. PMID 7720158
- [Background] Carlson JN, Crofts J, Walls RM, Brown CA 3rd. Direct Versus Video Laryngoscopy for Intubating Adult Patients with Gastrointestinal Bleeding. West J Emerg Med. 2015 Dec;16(7):1052-6. doi: 10.5811/westjem.2015.8.28045. Epub 2015 Dec 1. PMID 26759653
- [Background] Cortellazzi P, Caldiroli D, Byrne A, Sommariva A, Orena EF, Tramacere I. Defining and developing expertise in tracheal intubation using a GlideScope((R)) for anaesthetists with expertise in Macintosh direct laryngoscopy: an in-vivo longitudinal study. Anaesthesia. 2015 Mar;70(3):290-5. doi: 10.1111/anae.12878. Epub 2014 Oct 1. PMID 25271442
- [Background] Deutsch ES, Christenson T, Curry J, Hossain J, Zur K, Jacobs I. Multimodality education for airway endoscopy skill development. Ann Otol Rhinol Laryngol. 2009 Feb;118(2):81-6. doi: 10.1177/000348940911800201. PMID 19326756
- [Background] Griesdale DE, Liu D, McKinney J, Choi PT. Glidescope(R) video-laryngoscopy versus direct laryngoscopy for endotracheal intubation: a systematic review and meta-analysis. Can J Anaesth. 2012 Jan;59(1):41-52. doi: 10.1007/s12630-011-9620-5. Epub 2011 Nov 1. PMID 22042705
- [Background] Grundgeiger T, Roewer N, Grundgeiger J, Hurtienne J, Happel O. Body posture during simulated tracheal intubation: GlideScope((R)) videolaryngoscopy vs Macintosh direct laryngoscopy for novices and experts. Anaesthesia. 2015 Dec;70(12):1375-81. doi: 10.1111/anae.13190. Epub 2015 Sep 5. PMID 26342141
- [Background] Joffe AM, Aziz MF, Posner KL, Duggan LV, Mincer SL, Domino KB. Management of Difficult Tracheal Intubation: A Closed Claims Analysis. Anesthesiology. 2019 Oct;131(4):818-829. doi: 10.1097/ALN.0000000000002815. PMID 31584884
- [Background] Jones PM, Armstrong KP, Armstrong PM, Cherry RA, Harle CC, Hoogstra J, Turkstra TP. A comparison of glidescope videolaryngoscopy to direct laryngoscopy for nasotracheal intubation. Anesth Analg. 2008 Jul;107(1):144-8. doi: 10.1213/ane.0b013e31816d15c9. PMID 18635480
- [Background] Kennedy CC, Cannon EK, Warner DO, Cook DA. Advanced airway management simulation training in medical education: a systematic review and meta-analysis. Crit Care Med. 2014 Jan;42(1):169-78. doi: 10.1097/CCM.0b013e31829a721f. PMID 24220691
- [Background] Lewis SR, Butler AR, Parker J, Cook TM, Schofield-Robinson OJ, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adult patients requiring tracheal intubation: a Cochrane Systematic Review. Br J Anaesth. 2017 Sep 1;119(3):369-383. doi: 10.1093/bja/aex228. PMID 28969318
- [Background] Liu L, Tanigawa K, Kusunoki S, Tamura T, Ota K, Yamaga S, Kida Y, Otani T, Sadamori T, Takeda T, Iwasaki Y, Hirohashi N. Tracheal intubation of a difficult airway using Airway Scope, Airtraq, and Macintosh laryngoscope: a comparative manikin study of inexperienced personnel. Anesth Analg. 2010 Apr 1;110(4):1049-55. doi: 10.1213/ANE.0b013e3181d2aad7. PMID 20357149
- [Background] Liu TT, Li L, Wan L, Zhang CH, Yao WL. Videolaryngoscopy vs. Macintosh laryngoscopy for double-lumen tube intubation in thoracic surgery: a systematic review and meta-analysis. Anaesthesia. 2018 Aug;73(8):997-1007. doi: 10.1111/anae.14226. Epub 2018 Feb 6. PMID 29405258
- [Background] Martin LD, Mhyre JM, Shanks AM, Tremper KK, Kheterpal S. 3,423 emergency tracheal intubations at a university hospital: airway outcomes and complications. Anesthesiology. 2011 Jan;114(1):42-8. doi: 10.1097/ALN.0b013e318201c415. PMID 21150574
- [Background] Mosier JM, Stolz U, Chiu S, Sakles JC. Difficult airway management in the emergency department: GlideScope videolaryngoscopy compared to direct laryngoscopy. J Emerg Med. 2012 Jun;42(6):629-34. doi: 10.1016/j.jemermed.2011.06.007. Epub 2011 Sep 10. PMID 21911279
- [Background] Pieters BMA, Maas EHA, Knape JTA, van Zundert AAJ. Videolaryngoscopy vs. direct laryngoscopy use by experienced anaesthetists in patients with known difficult airways: a systematic review and meta-analysis. Anaesthesia. 2017 Dec;72(12):1532-1541. doi: 10.1111/anae.14057. Epub 2017 Sep 22. PMID 28940354
- [Background] Pieters BM, Wilbers NE, Huijzer M, Winkens B, van Zundert AA. Comparison of seven videolaryngoscopes with the Macintosh laryngoscope in manikins by experienced and novice personnel. Anaesthesia. 2016 May;71(5):556-64. doi: 10.1111/anae.13413. Epub 2016 Mar 12. PMID 26973253
- [Background] Pieters B, Maassen R, Van Eig E, Maathuis B, Van Den Dobbelsteen J, Van Zundert A. Indirect videolaryngoscopy using Macintosh blades in patients with non-anticipated difficult airways results in significantly lower forces exerted on teeth relative to classic direct laryngoscopy: a randomized crossover trial. Minerva Anestesiol. 2015 Aug;81(8):846-54. Epub 2014 Oct 14. PMID 25311949
- [Background] Platts-Mills TF, Campagne D, Chinnock B, Snowden B, Glickman LT, Hendey GW. A comparison of GlideScope video laryngoscopy versus direct laryngoscopy intubation in the emergency department. Acad Emerg Med. 2009 Sep;16(9):866-71. doi: 10.1111/j.1553-2712.2009.00492.x. Epub 2009 Aug 6. PMID 19664096
- [Background] Robitaille A, Williams SR, Tremblay MH, Guilbert F, Theriault M, Drolet P. Cervical spine motion during tracheal intubation with manual in-line stabilization: direct laryngoscopy versus GlideScope videolaryngoscopy. Anesth Analg. 2008 Mar;106(3):935-41, table of contents. doi: 10.1213/ane.0b013e318161769e. PMID 18292443
- [Background] Rothfield KP, Russo SG. Videolaryngoscopy: should it replace direct laryngoscopy? a pro-con debate. J Clin Anesth. 2012 Nov;24(7):593-7. doi: 10.1016/j.jclinane.2012.04.005. PMID 23101777
- [Background] Russell T, Khan S, Elman J, Katznelson R, Cooper RM. Measurement of forces applied during Macintosh direct laryngoscopy compared with GlideScope(R) videolaryngoscopy. Anaesthesia. 2012 Jun;67(6):626-31. doi: 10.1111/j.1365-2044.2012.07087.x. Epub 2012 Feb 21. PMID 22352799
- [Background] Sakles JC, Mosier J, Patanwala AE, Dicken J. Learning curves for direct laryngoscopy and GlideScope(R) video laryngoscopy in an emergency medicine residency. West J Emerg Med. 2014 Nov;15(7):930-7. doi: 10.5811/westjem.2014.9.23691. Epub 2014 Oct 29. PMID 25493156
- [Background] Waddington MS, Paech MJ, Kurowski IH, Reed CJ, Nicholls GJ, Guy DT, Day RE. The influence of gender and experience on intubation ability and technique: a manikin study. Anaesth Intensive Care. 2009 Sep;37(5):791-801. doi: 10.1177/0310057X0903700502. PMID 19775044
- [Background] Wetsch WA, Spelten O, Hellmich M, Carlitscheck M, Padosch SA, Lier H, Bottiger BW, Hinkelbein J. Comparison of different video laryngoscopes for emergency intubation in a standardized airway manikin with immobilized cervical spine by experienced anaesthetists. A randomized, controlled crossover trial. Resuscitation. 2012 Jun;83(6):740-5. doi: 10.1016/j.resuscitation.2011.11.024. Epub 2011 Dec 7. PMID 22155448